CLINICAL TRIAL: NCT03428282
Title: Effectiveness of Audio Visual Distraction Using Virtual Reality Eyeglasses Versus Tablet Device in Child Behavioral Management During Inferior Alveolar Nerve Block
Brief Title: Pain and Anxiety Control During Traditional Mandibular Anesthesia in Children Using Distracting Tools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Pedo-03-2017
Record Dates: First submitted 2017-12-26; First posted 2018-02-09 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Inferior Alveolar Nerve Block
MeSH Terms: interventions — Anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR Box (Experimental): Inferior alveolar nerve block will be performed with the aid of VR box as a means of distracting patients' attention.
  Interventions: Procedure: VR Box
- Tablet device (Experimental): Inferior alveolar nerve block will be performed with the aid of a tablet device as a means of distracting patients' attention.
  Interventions: Procedure: Tablet Device
- Anesthesia (Active Comparator): Inferior alveolar nerve block will be performed in the normal manner without any specific intervention to distract patients' attention. Classic anesthesia will be applied.
  Interventions: Drug: Anesthesia

INTERVENTIONS:
Procedure: VR Box — Distraction will be made during the injection of the drug using this method.
  Other Names: Virtual Reality Eyeglasses
  Arms: VR Box
Procedure: Tablet Device — Distraction will be made during the injection of the drug using this method
  Arms: Tablet device
Drug: Anesthesia — Anesthesia will be obtained by injecting the drug into the oral mucosa before performing the dental treatment.
  Arms: Anesthesia

SUMMARY:
The aim of this study is to evaluate the effectiveness of two different audiovisual distraction techniques (Audio Video eyeglasses "VR BOX"/ Tablet) in the management of anxious pediatric patients during inferior alveolar nerve block

Group A (Control group): IAN will be administrated with basic behavior guidance techniques and without using any type of distraction aids.

Group B: IAN will be administrated with using AV eyeglasses "VR BOX" and wireless headphone.

Group C: IAN will be administrated with using tablet device and wireless headphone

All of the children who experienced an inferior alveolar block with/without distraction will be assessed by using a combination of measures: Wong-Baker FACES (self-report), pulse rate (physiological) and behavior (using FLACC behavior rating scale "external evaluator

DETAILED DESCRIPTION:
This study will evaluate the effectiveness of two types of distraction aids that contain video using (tablet device or VR BOX eyeglasses) and audio distraction using wireless headphone. pain and anxiety will be evaluated during inferior alveolar nerve block using three behavioral scales, Wong-Baker FACES (self-report), pulse rate (physiological) and behavior (using FLACC behavior rating scale "external evaluator".

The first measure of heart pulse rate will be recorded directly when the patient seated comfortably on the dental chair, after anesthesia, the second heart pulse rate will be taken and the child patients will ask to choose a face that describe their status from one of the Wong Baker faces scale.

For each child patient, all of the body responses will be recorded during the whole procedure and then will be evaluated by an external assessor to determine the children behavioral score according to FLACC scale.

ELIGIBILITY:
Inclusion Criteria:

1. age between 6 and 10 years.
2. no previous dental experience.
3. definitely positive or positive ratings of Frank scale.
4. Need of IAN block for any dental treatment.

Exclusion Criteria:

1. previous dental experience
2. systematic or mental disorders.
3. definitely negative or negative ratings of Frankel scale
4. Any contraindication for regional anesthesia

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-02-10 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Pain levels | five minutes following the inferior alveolar nerve block injection.
  using self-reported Wong-Baker FACES pain scale with 0 indicating 'no pain' and five indicating 'worst pain'.
Anxiety levels | Within the first minute of injecting the needle into the oral mucosa (oral tissues).
  This will be evaluated using the Face-Legs-Activity-Cry-Consolability (FLACC) scale employing an external evaluator in which all of the body responses will be recorded once the needle penetrate the oral tissue.
  (0 low anxiety and pain level - 10 high anxiety and pain level)
Change in physiological pulse rate | (1) five minutes after the patient is seated comfortably on the dental chair, (2) five minutes following the injection of the anesthetic drug
  using Finger Pulse Oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Nour Al-Halabi, DDS, Principal Investigator — MSc student in Pedodontics, University of Damascus Dental School, Damascus, Syria; Zuhair AlNerabieah, DDS, Principal Investigator — MSc student in Pedodontics, University of Damascus Dental School, Syria; Nada Bshara, MD MSc Phd, Study Director — Associate Professor of Pedodontics, University of Damascus Dental School, Syria
Locations (1):
- Department of Peadodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madhok M, Teele M. Evaluation of nonpharmacologic methods of pain and anxiety management for laceration repair in the pediatric emergency department. Pediatrics. 2006 Sep;118(3):1321; author reply 1321-2. doi: 10.1542/peds.2006-1351. No abstract available. PMID 16951038
- [Background] Wang ZX, Sun LH, Chen AP. The efficacy of non-pharmacological methods of pain management in school-age children receiving venepuncture in a paediatric department: a randomized controlled trial of audiovisual distraction and routine psychological intervention. Swiss Med Wkly. 2008 Oct 4;138(39-40):579-84. doi: 10.4414/smw.2008.12224. PMID 18853287
- [Background] Al-Namankany A, Petrie A, Ashley P. Video modelling and reducing anxiety related to dental injections - a randomised clinical trial. Br Dent J. 2014 Jun;216(12):675-9. doi: 10.1038/sj.bdj.2014.497. PMID 24970519
- [Background] El-Sharkawi HF, El-Housseiny AA, Aly AM. Effectiveness of new distraction technique on pain associated with injection of local anesthesia for children. Pediatr Dent. 2012 Mar-Apr;34(2):e35-8. PMID 22583875
- [Background] Hoge MA, Howard MR, Wallace DP, Allen KD. Use of video eyewear to manage distress in children during restorative dental treatment. Pediatr Dent. 2012 Sep-Oct;34(5):378-82. PMID 23211912
- [Background] Fakhruddin KS, Hisham EB, Gorduysus MO. Effectiveness of audiovisual distraction eyewear and computerized delivery of anesthesia during pulp therapy of primary molars in phobic child patients. Eur J Dent. 2015 Oct-Dec;9(4):470-475. doi: 10.4103/1305-7456.172637. PMID 26929683